CLINICAL TRIAL: NCT04672005
Title: Modified FOLFIRINOX Alternated With Biweekly Gemcitabine Plus Nab-Paclitaxel in Untreated Metastatic Adenocarcinoma of the Pancreas
Brief Title: Modified FOLFIRINOX Alternated With Biweekly Gemcitabine Plus Nab-Paclitaxel Untreated Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lyudmyla Berim (Other)
Responsible Party: Sponsor-Investigator, Lyudmyla Berim, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020002395; 072011 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2020-11-09; First posted 2020-12-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Leucovorin; Irinotecan; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Regimen: mFOLFIRINOX + mGnabP (Experimental): All study participants will receive the following treatment:
  mFOLFIRINOX (28-day cycle)
  Day 1 and Day 15:
  Oxaliplatin 85 mg/m2 2-hour intravenous infusion followed by leucovorin 400 mg/m2 2-hour infusions with the addition of irinotecan 150 mg/m2 as a 90 minute infusion. 5-FU 2400 mg/m2 continuous intravenous infusion over 46 hours will follow irinotecan.
  Day 3 and Day 17:
  Pegylated-Granulocyte Colony Stimulating Facotr (peg-GCSF) 6 mg subcutaneous injection following disconnection of 5-FU infusion, first cycle and then per investigator discretion.
  Biweekly mGnabP (28-day cycle)
  Day 1 and Day 15:
  Nab-paclitaxel 125 mg/m2 infused over 30 minutes, immediately followed by Gemcitabine 1200 mg/m2 intravenously infused at the rate of 10mg/m2/min (over 120 minutes).
  Patients will receive one month of each regimen, alternately monthly until progression of disease.
  Interventions: Drug: Folfirinox alternating with Gemcitabine-nab-Paclitaxel

INTERVENTIONS:
Drug: Folfirinox alternating with Gemcitabine-nab-Paclitaxel — modified Folfirinox every 2 weeks and biweekly Gemcitabine plus Nab-Paclitaxel
  Other Names: Oxaliplatin; Leucovorin; Irinotecan; Nab-Paclitaxel; Gemcitabine

SUMMARY:
The main objective of the clinical trial is to determine if modified FOLFIRINOX (mFFX) alternated with biweekly Gemcitabine plus Nab-Paclitaxel (mGnabP) administered as a combined, front-line therapy will result in longer time to treatment failure (TTF) compared to the current standard of care with mFFX alone in treatment-naive patients with metastatic pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
1. Primary objective:

   To determine whether mFFX and mGnabP administered as a combined, alternating, front-line therapy can provide longer first line treatment for patients with metastatic pancreatic cancer, with the primary metric of time to treatment failure (TTF), including progression of disease (PD), death or treatment discontinuation due to toxicity.

   • Primary endpoint: TTF (treatment discontinuation due to toxicity, disease progression, or death).
2. Secondary objectives:

1) To determine objective response rate (ORR) of the regimen. 2) To determine progression-free survival (PFS) rate of the regimen. 3) To determine overall survival (OS) rate of the regimen. 4) To assess biomarker response (CA-19.9) to the regimen. 5) To examine safety and tolerability of the new regimen. 6) To examine health-related quality of life in patients receiving this regimen.

• Secondary endpoints:

1. ORR as determined by the proportion of subjects with either complete response (CR) or partial response (PR), as defined by RECIST 1.1.
2. PFS as determined by the time interval from the date of first dose of study regimen to first documented PD or death from any cause, whichever occurs first.
3. Overall survival (OS) as defined as the time interval from the date of the first dose of study regimen to date of death from any cause.
4. Biomarker response, measured by serum CA 19-9 levels every 4 weeks.
5. Safety and tolerability of the mFFX alternating with mGnabP regimen; Grade 3 and 4 toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Follow up for toxicity will be recorded for the first 30 days following the last chemotherapy cycle, and any long-term toxicity will be followed for up to 2 years after completion of study therapy.

3. Exploratory objectives:

1. To determine the tumor molecular profile prior to initiation of chemotherapy and correlate with treatment response.
2. To analyze ct-DNA as a biomarker of response to therapy and early detection of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed pancreatic adenocarcinoma.
2. Stage IV disease. The definitive diagnosis of metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data.
3. Subject must have received no prior therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed. If a subject received prior neoadjuvant or adjuvant chemotherapy, tumor recurrence must have occurred more than 6 months after completing the last dose of chemotherapy.
4. ECOG performance status of 0-1.
5. At least 18 years of age.
6. Evidence of measurable or non-measurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiotherapy.
7. Female patients of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male and female patients must agree to use effective barrier contraception during the period of therapy.
8. Adequate bone marrow function:

8a. ANC ≥ 1500/uL 8b.platelet count ≥ 100,000/uL 8c. hemoglobin ≥ 9.0 g/dL 9. Adequate hepatic function: 9a. Total bilirubin ≤ 1.5 X ULN 9b. AST (SGOT) ≤ 5 X ULN 9c. ALT (SGPT) ≤ 5 X ULN Patients with biliary obstruction must have restored biliary flow by placement of an endoscopic common bile duct stent or a percutaneous drainage.

10. Adequate renal function, Creatinine < 1.5x institutional ULN or calculated creatinine clearance ≥ 50 mL/min as estimated using the Cockcroft-Gault formula.

11. Partial thromboplastin time (PTT) < 1.2 x ULN and INR ≤ 1.5 x ULN, if not receiving anticoagulation therapy. For patients receiving anticoagulants, exceptions to these coagulation parameters are allowed if they are within the intended or expected range for their therapeutic use.

12. Subject must have no clinically significant abnormalities in urinalysis results (obtained ≤ 14 days prior to starting Cycle 1 Day 1).

13. Ability to understand the nature of this study protocol and give written informed consent. 14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Patients who meet any one of the following criteria will be excluded from this study.

1. Ineligible histology including non-adenocarcinomas, adenosquamous carcinoma, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct and ampullary carcinomas.
2. Any condition including the presence of laboratory abnormalities, which, in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study.
3. Presence of central nervous system metastases.
4. Life expectancy < 12 weeks.
5. Pregnancy (positive pregnancy test) or lactation.
6. Pre-existing sensory neuropathy > grade 1.
7. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
8. Major surgery without complete recovery in the past 4 weeks prior to screening.
9. Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.
10. Concurrent active infection.
11. Patient with uncontrolled and/ or active infection with HIV, Hepatitis B or Hepatitis C.
12. Patient who has a history of allergy or hypersensitivity to any of the study drugs.
13. Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, interstitial pulmonary fibrosis, pulmonary hypersensitivity pneumonitis.
14. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | 24 weeks
  The primary objective of this study is to determine time to treatment failure (TTF) in patients with metastatic pancreatic cancer treated in front line setting with mFOLFIRINOX (mFFX) alternating with biweekly Gemcitabine and nab-Paclitaxel (mGnabP).

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST 1.1 | 24 weeks
  Response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1 by independent radiology review) at 8 week intervals.
Progression-free survival (PFS) | 24 weeks
  To determine progression-free survival (PFS) rate of the regimen.
Overall survival (OS) | 24 weeks
  To determine overall survival (OS) rate of the regimen.
Safety and tolerability assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 24 weeks
  4. Safety and tolerability of the mFFX alternating with mGnabP regimen; Grade 3 and 4 toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Follow up for toxicity will be recorded for the first 30 days following the last chemotherapy cycle, and any long-term toxicity will be followed for up to 2 years after completion of study therapy.
EORTC QLQ-CIPN20 questionnaire | Administered at baseline prior to start of therapy, then every 8 weeks while receiving therapy, and at the end of treatment, average of 1 year
  Patient reported outcomes, examined through the EORTC QLQ-CIPN20 questionnaire
Correlation between variation in variant allele fraction (% cfDNA) or amplifications and tumor objective response during chemotherapy | Assessed at baseline prior to therapy, every 8 weeks interval through duration of therapy, and at end of treatment, average 1 year
  Correlation between variation in the variant allele fraction (% cfDNA) or amplifications and tumor objective response during chemotherapy

OTHER OUTCOMES:
Correlation between variation of ctDNA and progression free survival | 24 weeks
  Correlation between variation of ctDNA and progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmyla Berim, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (7):
- United States (7):
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health - Jersey City Medical Center, Jersey City, Jersey City, New Jersey
  - RWJBarnabas Health - Saint Barnabas Medical Center, Livingston, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No